CLINICAL TRIAL: NCT02542280
Title: Endometrial Injury May Increase the Pregnancy Rate in Patients Undergoing Intrauterine Insemination
Brief Title: Does Endometrial Injury Improve Intrauterine Insemination Outcome?
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Bahaa Eldin Ahmed, lesturer in Obstetrics and Gynecology., Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: abahaa050301
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Results first posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2015-11

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Insemination, Artificial; Ovulation Induction

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- endometrial injury (Experimental): Endometrial injury during ovarian stimulation combined with intrauterine insemination.
  Interventions: Procedure: endometrial injury.; Procedure: intrauterine insemination; Drug: ovarian stimulation
- no endometrial injury (Active Comparator): Ovarian stimulation combined with intrauterine insemination.
  Interventions: Procedure: intrauterine insemination; Drug: ovarian stimulation

INTERVENTIONS:
Procedure: endometrial injury. — Endometrial injury using a pipelle biopsy catheter on day (5, 6 or 7) of the stimulation cycle combined with the intrauterine insemination.
  Other Names: endometrial scratch.; endometrial sample.
  Arms: endometrial injury
Procedure: intrauterine insemination — Placement of washed sperm in the uterus using a catheter, around the time of ovulation.
  Other Names: artificial insemination
Drug: ovarian stimulation — Inducing ovulation by human menopausal gonadotrophin ampoules given intramuscular starting from cycle day two, till the leading follicle reaches 16 - 18 mm.
  Other Names: controlled ovarian hyperstimulatiom

SUMMARY:
The investigator suggests that local endometrial injury using pipelle catheter performed in the follicular phase (cycle day 5, 6 or 7) of the stimulation cycle may improve the pregnancy rates among patients undergoing intrauterine insemination.

DETAILED DESCRIPTION:
In a selected group of patients with repeated implantation failure, endometrial injury in the preceding cycle may improve ICSI outcome.

Little is known about the efficacy of this procedure in improving intrauterine insemination outcome.

Also little is known about the effect of this procedure if done in the stimulation cycle weather in ICSI or intrauterine insemination cycles.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 38 years.
* patent fallopian tunes.
* mild male factor.
* anovulation.
* unexplained infertility.

Exclusion Criteria:

* indications for ICSI.
* evidence of pelvic inflammatory disease.

Ages: 18 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 360 (Actual)
Dates: Start 2013-07; Primary Completion 2015-07 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Bahaa, Principal Investigator — Lecturer in Obstetrics and Gynecology, faculty of medicine, Ain Shams University.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the infertility clinic and given appointments to go to the Assisted Reproductive Technology unit to start the process of IUI.
Pre-assignment Details: 11 patients were excluded because they did not show up for their appointments in assisted reproductive technology unit.
Groups:
- Endometrial Injury: Endometrial injury during ovarian stimulation cycle combined with intrauterine insemination.
  endometrial injury: Endometrial injury using a pipelle biopsy catheter on day (5, 6 or 7) of the stimulation cycle combined with the intrauterine insemination.
  intrauterine insemination: Placement of washed sperm in the uterus using a catheter, around the time of ovulation.
  ovarian stimulation: Inducing ovulation by clomiphene citrate 100mg orally (from cycle day 2 for 5 days) and human menopausal gonadotrophin ampoules given intramuscular starting from cycle day two, till the leading follicle reaches 16 - 18 mm.
- no Endometrial Injury: Ovarian stimulation combined with intrauterine insemination.
  intrauterine insemination: Placement of washed sperm in the uterus using a catheter, around the time of ovulation.
  ovarian stimulation: Inducing ovulation by clomiphene citrate 100mg orally (from cycle day 2 for 5 days) and human menopausal gonadotrophin ampoules given intramuscular starting from cycle day two, till the leading follicle reaches 16 - 18 mm.
Period: Overall Study
Arm/Group | Endometrial Injury | no Endometrial Injury
Started | 174 | 175
Completed | 162 | 167
Not Completed | 12 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Endometrial Injury | no Endometrial Injury | Total
Number analyzed (Participants) | 162 | 167 | 329
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.57 (3.99) | 29.52 (4.09) | 29.1 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162 | 167 | 329
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Egypt | 162 | 167 | 329
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.5 (4) | 29.35 (3.02) | 28.9 (3.6)

OUTCOME MEASURES:

1. Primary Outcome: Chemical Pregnancy Rate
Description: Human chorionic gonadotrophin (b-hcg) detection in serum two weeks after intrauterine insemination.
Time Frame: two weeks after intrauterine insemination
Measure: Number; unit: participants
Arm/Group | Endometrial Injury | no Endometrial Injury
Number analyzed (Participants) | 162 | 167
participants | 40 | 19

2. Primary Outcome: Clinical Pregnancy Rate
Description: Ultrasound detection of an intrauterine positive fetal heart pulsations
Time Frame: six weeks
Measure: Number; unit: participants
Arm/Group | Endometrial Injury | no Endometrial Injury
Number analyzed (Participants) | 162 | 167
participants | 32 | 13

ADVERSE EVENTS:
Arm/Group | Endometrial Injury | no Endometrial Injury
Serious Adverse Events (participants affected / at risk) | 0/162 | 0/167
Other Adverse Events (participants affected / at risk) | 0/162 | 0/167

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No